CLINICAL TRIAL: NCT05962580
Title: of Anterior Cruciate Ligament Reconstruction With and Without Lateral Extra-Articular Tenodesis Between High Demand Patients: Randomized Controlled Trial
Brief Title: Anterior Cruciate Ligament Reconstruction With and Without Lateral Extra-Articular Tenodesis Among High Demand Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD 13/2021
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Anterior Cruciate Ligament Tear
Keywords: anterior cruciate ligament tear; anterolateral instability; retear; extra articular tenodesis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolated anterior cruciate ligament recnostruction with lateral extra articular tenodesis (Experimental): Arthroscopic anatomical single bundle anterior cruciate ligament reconstruction with modified Lemiere technique for extra-articular tenodesis
  Interventions: Procedure: Isolated anterior cruciate ligament reconstruction with lateral extra articular tenodesis
- Isolated anterior cruciate ligament recnostruction without lateral extra articular tenodesis (Active Comparator): Arthroscopic anatomical single bundle anterior cruciate ligament reconstruction only
  Interventions: Procedure: Isolated anterior cruciate ligament reconstruction only

INTERVENTIONS:
Procedure: Isolated anterior cruciate ligament reconstruction with lateral extra articular tenodesis — Anatomical single bundle ACLR with modified Lemiere technique
  Arms: Isolated anterior cruciate ligament recnostruction with lateral extra articular tenodesis
Procedure: Isolated anterior cruciate ligament reconstruction only — arthroscopic anatomical single bundle ACL Reconstruction
  Arms: Isolated anterior cruciate ligament recnostruction without lateral extra articular tenodesis

SUMMARY:
Anterior Cruciate Ligament Reconstruction with and without Lateral Extra-Articular Tenodesis between high demand patients

DETAILED DESCRIPTION:
It is a randomized control trial comparing between isolated anterior cruciate ligament reconstruction with and without lateral extra articular tenodesis between high demand and high risk groups with high pivot regarding failure rate (primary out come) and patient reported functions score (IKDC and Lysholm)

ELIGIBILITY:
Inclusion Criteria:

* High demand patients (manual workers, athletes,...etc.).
* Normal average body mass index ( 18.5 - 24.9 ).
* Age <40 years old.
* Patients will be diagnosed as ACL tear by the following:

  1. History of knee traumatic event.
  2. Clinical examination ( positive Lachman test and pivot shift test).
  3. Radiological evidence of ACL tear by MRI.
* patient with high pivot shift test.

Exclusion Criteria:

* Generalized ligamentous laxity.
* Other intra or extra articular knee injuries.
* Previous ACL surgery on the affected knee.
* Bilateral ACL injuries.
* Significant Articular surface injury.
* Medical comorbidities
* Patients with malalignment ( genu varum, genu valgum or genu recurvatum )
* Neuromuscular disorders
* Knee arthritic changes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
failure rate | one year follow up
  retear of ACL graft confirmed by clinical examination and MRI

SECONDARY OUTCOMES:
International knee documentation committee score (IKDC) | at 3,6,9,12 months
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)
Lysholm score | at 3,6,9,12 months
  The Lysholm Knee Score calculates and grades an overall score from 0 to 100 based on 8 domains: squatting, locking, pain, stair climbing, support, instability, and edema. Physicians use this condition-specific, subjective outcome score to assess patient progress after surgery or injury to the knee. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)
antero-posterior instability measure | at 3,6,9 and 12 months
  measure AP instability by KT1000 lachmeter for injured and non injured knee
side to side KT 1000 lachmeter difference | one year follow up
  measure side to side KT 1000 lachmeter difference by (injured - noninjured)

CONTACTS AND LOCATIONS:
Overall Officials: Amr Mo Abdelhady, Professor, Study Chair — Faculty of medecine, Ain shams university; Mohamed Ha Sobhey, Professor, Study Director — Faculty of medecine, Ain shams university; Moustapha Al ElAbd, lecturer, Study Director — Faculty of medecine, Ain shams university; Yehia Mo Haroun, Lecturer, Study Director — Faculty of medecine, Ain shams university; Ahmed Ab Amer, Msc, Principal Investigator — Faculty of medecine, Ain shams university
Locations (1):
- Ahmed Abdel Salam Abdel Halim, Cairo, Abbasia, Egypt